CLINICAL TRIAL: NCT07163299
Title: Selective Intra-arterial Hypothermic Magnesium Sulfate Infusion in Combination With Endovascular Thrombectomy in Acute Ischemic Stroke: A Phase 1/2 Randomized Clinical Trial
Brief Title: Intra-arterial Selective Hypothermic Magnesium Sulfate Infusion in Combination With Endovascular Thrombectomy in Acute Ischemic Stroke
Acronym: ICE-MAG
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor of Neurology, Xuanwu Hospital, Capital Medical University, Capital Medical University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ICE-MAG
Record Dates: First submitted 2025-08-27; First posted 2025-09-09 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Acute Ischemic Stroke
Keywords: thrombectomy; magnesium sulfate; intra-arterial hypothermic
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: This study was divided into two parts. The first part was a dose escalation study (non-randomized) using a "3+3" design. The second part was a randomized, parallel, open-label, endpoint-blinded study conducted at the maximum tolerated dose (MTD)
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Selective intra-arterial hypothermic magnesium sulfate infusion of low volume (Experimental): Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (350 ml).
  Interventions: Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (350 ml).
- Selective intra-arterial hypothermic magnesium sulfate infusion of moderate volume (Experimental): Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (500 ml).
  Interventions: Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (500 ml).
- Selective intra-arterial hypothermic magnesium sulfate infusion of high volumn (Experimental): Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (650 ml).
  Interventions: Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (650 ml).
- Control (Sham Comparator): Endovascular thrombectomy alone
  Interventions: Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (350 ml).; Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (650 ml).

INTERVENTIONS:
Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (350 ml). — According to patient's weight, magnesium sulfate (MgSO4) will be diluted to 350 ml 4°C saline solution (0.6μmol/kg/ml). During the thrombectomy procedure, a micro-catheter will be advanced until it reaches beyond the clot responsible for the ischemic symptoms, then cold 50 ml MgSO4 solution will be infused into the ischemic territory at 10 ml/min through the micro-catheter. After that, thrombectomy with a stent retriever will be performed to recanalize the occluded vessel as soon as possible. Immediately after successful thrombectomy, cold MgSO4 solution will be re-infused into the ischemic brain tissue through the catheter at a rate of 30 ml/min for 10 min.
  Arms: Control; Selective intra-arterial hypothermic magnesium sulfate infusion of low volume
Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (500 ml). — According to patient's weight, magnesium sulfate (MgSO4) will be diluted to 500 ml 4°C saline solution (0.6μmol/kg/ml). During the thrombectomy procedure, a micro-catheter will be advanced until it reaches beyond the clot responsible for the ischemic symptoms, then cold 50 ml MgSO4 solution will be infused into the ischemic territory at 10 ml/min through the micro-catheter. After that, thrombectomy with a stent retriever will be performed to recanalize the occluded vessel as soon as possible. Immediately after successful thrombectomy, cold MgSO4 solution will be re-infused into the ischemic brain tissue through the catheter at a rate of 30 ml/min for 10 min. Then pause for 5 min, followed by another 5 min of infusion at the original rate.
  Arms: Selective intra-arterial hypothermic magnesium sulfate infusion of moderate volume
Procedure: Endovascular thrombectomy combination with selective intra-arterial hypothermic magnesium sulfate infusion (650 ml). — According to patient's weight, magnesium sulfate (MgSO4) will be diluted to 650 ml 4°C saline solution (0.6μmol/kg/ml). During the thrombectomy procedure, a micro-catheter will be advanced until it reaches beyond the clot responsible for the ischemic symptoms, then cold 50 ml MgSO4 solution will be infused into the ischemic territory at 10 ml/min through the micro-catheter. After that, thrombectomy with a stent retriever will be performed to recanalize the occluded vessel as soon as possible. Immediately after successful thrombectomy, cold MgSO4 solution will be re-infused into the ischemic brain tissue through the catheter at a rate of 30 ml/min for 10 min. Then pause for 5 min, followed by intermittent infusion at the original rate for another 5 min twice. The interval between two times is also 5 min.
  Arms: Control; Selective intra-arterial hypothermic magnesium sulfate infusion of high volumn

SUMMARY:
The primary objective of this study is to estimate the safety and effectiveness of selective intra-arterial hypothermic magnesium sulfate infusion after endovascular thrombectomy in patients with acute ischemic stroke

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-80 years old (including critical value);
2. No gender restrictions;
3. The clinical diagnosis is acute ischemic stroke of the anterior circulation, and the site of acute occlusion of the responsible vessel is located in the intracranial segment of the internal carotid artery and the M1 or M2 segment of the middle cerebral artery;
4. The symptoms and signs are consistent with acute anterior circulation ischemic stroke, NIHSS≥6;
5. The time from onset to endovascular thrombectomy of acute ischemic stroke is within 24 hours;
6. Indications for endovascular thrombectomy of acute ischemic stroke: ① ASPECTS score ≥ 6 points, within 6 hours of onset; ② 6-16 hours after onset, meeting DEFUSE-3 criteria (infarct core volume < 70 mL, mismatch rate ≥ 1.8 and mismatch volume > 15 mL) or DAWN criteria (NIHSS ≥ 10 and infarct core volume < 31 mL); Or NIHSS ≥ 20 and infarct volume 31-51 mL); ③ Within 16-24 hours of onset, meet DAWN criteria (NIHSS ≥ 10 points and infarct core volume < 31mL); Or NIHSS ≥ 20 points and infarct volume 31-51 mL)
7. The mRS score before stroke is 0-1 points;
8. Written informed consent provided by the patients or their legal relatives.

Exclusion Criteria:

General exclusion criteria:

1. Clinical manifestations suggest the presence of intracranial cerebral parenchymal hemorrhage or subarachnoid hemorrhage (even if imaging results are normal);
2. During a stroke, accompanied by epilepsy, an accurate NIHSS score cannot be obtained;
3. Accompanied by coma or mental disorders, it may interfere with the assessment of neurological function;
4. History of allergy to iodinated contrast agents or history of anaphylactic shock;
5. Baseline blood glucose<50mg/dL (2.78mmol) or>400mg/dL (22.20mmol);

   *Acceptable fingertip blood glucose results
6. Baseline platelet count<50 × 10^9/L;
7. Recently (i.e. within 30 days prior to inclusion in the study), there has been a history of significant gastrointestinal or other clinically significant bleeding; Active bleeding, abnormal coagulation factors, or bleeding tendency (taking anticoagulant drugs with INR ≥ 3 or PT ≥ 3 × ULN; if the researcher believes that the subject has no coagulation dysfunction, there is no need to wait for coagulation test results to determine whether to enroll);
8. During a stroke, there may be fever or active infections that require systemic treatment (such as active pulmonary tuberculosis);
9. History of chronic heart failure with NYHA criteria>1; Uncontrolled hypertension (systolic blood pressure>180mmHg or diastolic blood pressure>105mmHg after standardized treatment), hypotension (systolic blood pressure ≤ 100mmHg after standardized treatment), unstable angina, myocardial infarction, or bypass or stent surgery within 6 months;
10. Accompanied by pulmonary diseases such as chronic obstructive pulmonary disease, tuberculosis, pneumonia, pneumothorax, atelectasis, pulmonary fibrosis, bronchopulmonary dysplasia, pleural effusion, acute respiratory distress syndrome, irregular breathing, etc;
11. Severe liver and kidney dysfunction, including but not limited to: cirrhosis, hepatic encephalopathy, ascites, renal failure or uremia (Ccr<25ml/min), hepatorenal syndrome, etc;
12. Pregnant or lactating women;
13. Patients with acute stroke within 48 hours after percutaneous cardiovascular and cerebrovascular intervention and major surgery;
14. Currently participating in interventional clinical trials and using research drugs or medical devices;
15. Participants may not be able to complete this study due to other reasons or may not be considered eligible for inclusion by the researchers;

Image exclusion criteria:

1. CTA/MRA/DSA shows excessive vessel curvature, which may hinder the delivery of interventional instruments;
2. Suspected cerebral vasculitis based on medical history and CTA/MRA/DSA;
3. Suspected aortic dissection based on medical history and CTA/MRA/DSA;
4. CTA/MRA/DSA confirmed multi vessel regional occlusion (such as bilateral anterior circulation or anterior/posterior circulation, extracranial carotid artery with intracranial tandem lesions), or clinical evidence of bilateral infarction or multi regional infarction;
5. CTA/MRA/DSA confirms moyamoya disease or moyamoya syndrome;
6. CT/MRI confirms significant effect of midline shift;
7. CT/MRI confirms the presence of intracranial tumors (excluding small meningiomas);
8. CT/MRI confirms the presence of intracranial hemorrhage.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
Mortality at 90 days | 90 days after intra-arterial hypothermic magnesium sulfate infusion
Effectiveness evaluation indicators: | 90 days after intra-arterial hypothermic magnesium sulfate infusion
  Percentage of subjects with 90 days of functional independence (defined as mRS 0-2) (%) Evaluation time: 90 d (±14 d) after surgery

SECONDARY OUTCOMES:
Grade 3-5 Treatment Emergent Adverse Event (TEAE) related to intervention occurring during treatment period | Within 72 hours after intra-arterial hypothermic magnesium sulfate infusion
  TEAE includes but not limited to cardiovascular system response, abnormal electrocardiogram, water-electrolyte imbalance, core temperature decreasing, vascular spasm, shiver, infect, disturbance of consciousness.
All Treatment Emergent Adverse Event (TEAE) related to intervention occurring during treatment period | Within 72 hours after intra-arterial hypothermic magnesium sulfate infusion
All Treatment Emergent Adverse Event (TEAE) occurring during treatment period | Within 72 hours after intra-arterial hypothermic magnesium sulfate infusion
The proportion of symptomatic/asymptomatic intracranial hemorrhage within 24 hours | Within 24 hours after intra-arterial hypothermic magnesium sulfate infusion
No reflux rate | 24 hours (±6 hours) after surgery
  No reflux rate, defined as the percentage of subjects with a decrease in CBV or CBF by more than 15% compared to the contralateral side at 24 hours after treatment (%)

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China